CLINICAL TRIAL: NCT00632372
Title: CRT-D Based Heart Failure Monitoring Study
Brief Title: Cardiac Resynchronization Therapy (CRT) Based Heart Failure Monitoring Study
Acronym: zLAP
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 60015786
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- HeartPOD™ System with Cardiac Resynchronization Therapy: All patients will receive both a HeartPod device and a CRT-D device.
  Interventions: Device: Cardiac Resynchronization Therapy; Device: HeartPOD™ System

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy — Pacing of the left ventricle to resynchronize ventricular contraction.
  Other Names: CRT-D
Device: HeartPOD™ System — Left atrial pressure monitoring.

SUMMARY:
The purpose of this study is to collect and analyze electrical measurements, timing, and signals from a CRT-D device in heart failure patients who either already have an implanted left atrial pressure sensor or will undergo a simultaneous implantation of a left atrial pressure sensor and a CRT-D device. These devices may be placed at the same time or separately (staged procedure) at the discretion of the investigator. A comparison will be made between the information gathered from the CRT-D system and the information gathered by the left atrial pressure sensor.

DETAILED DESCRIPTION:
This is a multi-center feasibility study.

.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and ≤ 85.
* Have an approved indication per ACC/AHA/HRS guidelines for implantation of a CRT-D. Alternatively, the patient may already have in place an existing Promote CRT-D or other SJM CRT device with similar functions, or have a CRT-D device that requires a generator change. In addition, the patient may be already enrolled in HOMEOSTASIS I or II and completed the 12-month follow-up.
* Central venous vascular access.
* Have a legally marketed right atrial bipolar pacing lead, a right ventricular bipolar defibrillation lead, and a left ventricular bipolar pacing lead.
* Demonstrate capability of Valsalva maneuver with airway pressure > 40 mm Hg for ≥10 seconds.
* The subject and the treating physician agree that the subject is geographically stable and willing to comply with all required post-procedure follow-up, and that the patient is capable of correct device use as outlined in the protocol.
* The subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board or Ethics Committee of the respective clinical site

Exclusion Criteria:

* Intractable HF with resting symptoms despite maximal medical therapy (AHA/ACC Stage D) or active listing for cardiac transplantation (<6 months survival expected).
* Resting systolic blood pressure < 90 or > 180 mm Hg.
* Acute Myocardial Infarction (MI), unstable ischemic syndrome within the last 6 weeks.
* Percutaneous coronary intervention (PCI) or cardiac surgery performed or planned within ± 6 weeks.
* Coexisting stenotic valve lesions, vegetations, hypertrophic cardiomyopathy, amyloidosis or other infiltrative heart disease, constrictive, restrictive disease, tamponade, or moderate or large pericardial effusion.
* Subject has a history of deep venous thrombosis or pulmonary embolism within the last 6 months.
* Surgical correction of congenital heart disease involving atrial septum that will prevent safe implantation of the SJM HeartPOD ISL.
* Cerebral Vascular Accident (CVA) or Transient Ischemic Attacks (TIA's) within the last 6 months. History of uncorrected cerebral vascular disease.
* Atrial or ventricular thrombus, tumor or systemic thromboembolism.
* Atrial septal defect or clinically significant patent foramen ovale.
* Life expectancy less than one year from malignancy, primary pulmonary hypertension, renal, hepatic, or neurological condition, etc.
* Gastrointestinal bleeding during the last 6 months.
* Coagulopathy or uninterruptible anticoagulation therapy or unable to take antiplatelet medications.
* Creatinine > 2.4 gm/dl (212 µmol/L) at enrollment.
* Active systemic infection.
* The subject is currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
* Have a contraindication for an emergency thoracotomy
* Have a hypersensitivity to a single 1.0mg dose of dexamethasone sodium phosphate or short term contact with heparin.
* Positive pregnancy test at enrollment or planning a pregnancy in the next 12 months.
* Patient is pacemaker dependent, where cessation of pacemaker function consistently results in syncope or ventricular asystole.
* Incompatible previously implanted intracardiac devices.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with class III heart failure and a CRT-D device implanted.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determine which heart failure monitoring feature acquired by the CRT device correlates most closely with simultaneously measured left ventricular filling pressure, as measured by left atrial pressure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Troughton, MD, Principal Investigator — Christchurch Hospital - Christchurch, New Zealand
Locations (10):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Sanger Clinic, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Medical Univserity of South Carolina, Charleston, South Carolina
- Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan WY, Blomqvist A, Melton IC, Noren K, Crozier IG, Benser ME, Eigler NL, Gutfinger D, Troughton RW. Effects of AV delay and VV delay on left atrial pressure and waveform in ambulant heart failure patients: insights into CRT optimization. Pacing Clin Electrophysiol. 2014 Jul;37(7):810-9. doi: 10.1111/pace.12362. Epub 2014 Feb 6. PMID 24502608